CLINICAL TRIAL: NCT07302568
Title: The Effects of Exercise and Gezaixi (Taiwanese Opera) Interventions on Community-Dwelling Older Adults
Brief Title: Exercise and Gezaixi Interventions on Community-Dwelling Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wu Gueyhau, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202503em021
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Functional Decline; Community-Dwelling Older Adults
Keywords: Exercise; Gezaixi (Taiwanese Opera); Resistance Exercise; Strength Training; Community-Dwelling Older Adults
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Resistance Training; Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise with Taiwanese Opera Elements (Experimental): Weekly 2-hour group sessions for 12 consecutive weeks; 60 minutes progressive strength training plus 60 minutes Taiwanese opera-based activities.
  Interventions: Behavioral: Strength Training plus Taiwanese Opera-based Activities
- Usual Activity (No Intervention): Control : Usual Activity（No Intervention）

INTERVENTIONS:
Behavioral: Strength Training plus Taiwanese Opera-based Activities — Group-based exercise delivered at community centers for community-dwelling adults aged ≥65 years. Frequency: once per week. Session length: 120 minutes per session (60 minutes progressive strength training + 60 minutes Taiwanese opera-based activities integrating singing, reciting, acting, and martial arts). Total duration: 12 consecutive weeks.
  * Content and progression: Strength training targets major muscle groups (e.g., sit-to-stand, rowing/pulling with elastic bands, hip abduction, calf raises) using body weight, elastic bands, or light dumbbells; intensity targeted at moderate level (Borg RPE 11-13) and progressed by resistance/repetitions as tolerated. The opera-based segment includes rhythmic movement, balance drills, upper-/lower-limb coordination, posture and breathing, and simple choreographed sequences adapted from Taiwanese opera elements. Each session includes ~10 minutes warm-up and ~10 minutes cool-down with flexibility and breathing exercises. Approximate group size:
  Other Names: Opera-integrated Exercise Program for Older Adults
  Arms: Exercise with Taiwanese Opera Elements

SUMMARY:
This interventional study evaluates a 12-week, once-weekly group exercise program combining 60 minutes of progressive strength training and 60 minutes of Taiwanese opera-based activities for community-dwelling adults aged ≥65 in Taipei. The primary aim is to delay frailty and functional decline by improving physical fitness and independence. Primary outcomes are muscle strength, calf circumference, and SOF frailty score; secondary outcomes are BSRS-5, GGDS-5, and SARC-F. The study uses a non-randomized, parallel two-arm design (exercise vs. usual activity), open-label, with assessments at baseline and week 12.

DETAILED DESCRIPTION:
Participants attend weekly 120-minute sessions for 12 consecutive weeks at community centers. Strength training targets major muscle groups using body weight, elastic bands, or light dumbbells at moderate intensity (Borg RPE 11-13) with progressive overload. The Taiwanese opera-based segment integrates singing, reciting, acting, and martial arts elements to promote balance, coordination, posture, and endurance. Sessions include warm-up and cool-down. Certified C-level instructors lead classes; adherence and adverse events are monitored each session. Statistical analysis will compare pre-post changes within groups (paired t-tests) and between-group differences in change scores (independent t-tests or ANCOVA adjusting for baseline values). Missing data will be handled primarily using complete case analysis, with sensitivity analyses using linear mixed-effects models under a MAR assumption or multiple imputation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years.
* Community-dwelling older adults residing in Taipei.
* Able to ambulate independently (with or without assistive device).
* Able to communicate and provide informed consent.

Exclusion Criteria:

* Unstable cardiopulmonary disease or uncontrolled hypertension.
* Severe cognitive impairment affecting participation.
* Recent major surgery or fracture within the past 3 months.
* Any contraindication to moderate-intensity exercise as assessed by the study team.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | From enrollment to the end of intervention at 12 week
  Change in muscle strength from baseline to week 12, measured using standardized tests (e.g., handgrip strength with a dynamometer in kilograms, or 30-second chair stand repetitions). Higher values indicate better strength.
Calf Circumference | rom enrollment to the end of treatment at 12 weeks
  Change in calf circumference (centimeters) measured at the widest point of the non-dominant calf using a non-stretchable tape. Larger circumference generally indicates better muscle mass.
Study of Osteoporotic Fractures (SOF) frailty score | From enrollment to the end of treatment at 12 week
  Change in Study of Osteoporotic Fractures (SOF) frailty score (range 0-3; higher scores indicate greater frailty)

SECONDARY OUTCOMES:
Brief Symptom Rating Scale 5-item (BSRS-5) | From enrollment to the end of treatment at 12 weeks
  Change in the total score on the 5-item Brief Symptom Rating Scale (BSRS-5); higher scores indicate greater psychological distress. Scores range from 0 to 20.
Geriatric Depression Scale score 5-item(GGDS-5) | From enrollment to the end of treatment at 12 weeks
  Change in the 5-item Geriatric Depression Scale (GDS-5) score; higher scores indicate more depressive symptoms. Scores range from 0 to 5.
SARC-F | From enrollment to the end of treatment at 12 weeks
  Description: Change in SARC-F questionnaire score for sarcopenia risk (range 0-10; higher scores indicate higher risk).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taitau District, Taiwan

IPD SHARING:
Plan to Share IPD: No